CLINICAL TRIAL: NCT00003123
Title: A Phase II Trial of Ethyol (Amifostine) in Adult Patients With Advanced Myelodysplastic Syndromes
Brief Title: Amifostine in Treating Patients With Advanced Myelodysplastic Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Providence Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065882; PH-890; ALZA-97-018-ii; NCI-V97-1350
Record Dates: First submitted 1999-11-01; First posted 2004-08-12 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2004-01

CONDITIONS: Myelodysplastic Syndromes
Keywords: refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts | interventions — Amifostine

INTERVENTIONS:
Drug: amifostine trihydrate

SUMMARY:
RATIONALE: Amifostine may be effective in helping blood counts return to normal in treating patients with myelodysplastic syndrome.

PURPOSE: Phase II trial to study the effectiveness of amifostine in treating patients with advanced myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the overall hematologic response rate to amifostine in patients with advanced myelodysplastic syndrome. II. Determine the toxic effects of amifostine in these patients.

OUTLINE: This is an open label study. Patients receive intravenous amifostine over 15 minutes three times a week. Patients failing to respond by 8 weeks undergo dose escalation. Nonresponding patients are removed from the study by 12 weeks. Therapy is continued for up to six months in responding patients. Patients are observed for duration of response upon therapy discontinuation. Patients who relapse will have therapy resumed at the previous dose. Patients will be followed until death.

PROJECTED ACCRUAL: A maximum of 36 patients will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven advanced myelodysplastic syndrome (MDS), including: Refractory anemia Refractory anemia with ringed sideroblasts Refractory anemia with excess blasts Refractory anemia with excess blasts in transformation MDS with at least bicytopenia No chronic myelomonocytic leukemia No acute leukemia

PATIENT CHARACTERISTICS: Age: 17 and over Performance Status: ECOG 0-2 Life Expectancy: Greater than 6 months Hematopoietic: Hemoglobin less than 8.5 g/dL Absolute granulocyte count less than 1,000 g/dL Platelet count less than 70,000/mm3 Hepatic: No major hepatic problems Renal: No major renal problems Cardiovascular: No major cardiac disease Other: Prior transfusion of blood products is allowed Not pregnant Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior cytokine therapy is allowed Chemotherapy: No prior chemotherapy Endocrine therapy: Prior steroid therapy is allowed Radiotherapy: Not specified Surgery: Not specified Other: Prior leucovorin calcium and pyridoxine allowed

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 1997-08

CONTACTS AND LOCATIONS:
Overall Officials: Howard R. Terebelo, DO, Study Chair — Providence Hospital
Locations (7):
- United States (7):
  - Osteopathic Medical Oncology and Hematology, P.C., Clinton Township, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Garden City Hospital, Garden City, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - Providence Hospital Cancer Center, Southfield, Michigan
  - Cleveland Clinic Cancer Center, Cleveland, Ohio

REFERENCES:
- [Result] Terebelo H, Marsico D, Shurafa M, et al.: A phase II trial of amifostine in patients with advanced myelodysplastic syndromes. [Abstract] Proceedings of the American Society of Clinical Oncology 18: A82, 23a, 1999.